CLINICAL TRIAL: NCT03819660
Title: Long Term Safety Study of Amifampridine Phosphate in Ambulatory Patients With Spinal Muscular Atrophy (SMA) Type 3
Brief Title: Long Term Safety of Amifampridine Phosphate in Spinal Muscular Atrophy 3
Acronym: SMA3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of indication not being pursued
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-002
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Spinal Muscular Atrophy Type 3
Keywords: Type 3
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Amifampridine; Tablets

STUDY DESIGN:
Intervention Model Description: Open-label, extension study , long term safety and tolerability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- amifampridine phosphate (Experimental): The dose of amifampridine was based on optimal neuromuscular benefit determined from the Run-in Period from SMA-001 or could be modified as the discretion of the Investigator. The maximum single dose was 20 mg. The dose range for patients 6 to 16 years of age was 15 to 60 mg, and for those 17 years and older the range was from 30 to 80 mg daily.
  Interventions: Drug: Amifampridine Phosphate 10 MG Oral Tablet

INTERVENTIONS:
Drug: Amifampridine Phosphate 10 MG Oral Tablet — Oral tablets

SUMMARY:
A long term safety study of amifampridine phosphate in patients with spinal muscular atrophy (SMA) Type 3.

DETAILED DESCRIPTION:
This open-label outpatient extension study was designed to evaluate the long-term safety and tolerability of amifampridine in patients diagnosed with SMA Type 3. In addition, the evaluation of the effects of amifampridine on the QoL was performed. The study was planned to enroll those patients who had completed the SMA-001 study and after all final evaluations for that study had been completed, or those who demonstrated benefit after completing the dose titration period but failed to meet the randomization criteria on Day 0 of SMA-001.

The duration of participation for each patient was expected to be at least 12 months as patients could continue in the study until amifampridine was approved by Regulatory Agencies or the clinical development of amifampridine was terminated for this indication. In addition to amifampridine, patients continued to receive previous concomitant medications, as needed.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in this study must meet all the following inclusion criteria:

1. Participated in the SMA-001 study
2. Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.
3. Female patients of childbearing potential must have a negative pregnancy test (urine human chorionic gonadotropin [HCG] at the end of SMA-001 study); and must practice an effective, reliable contraceptive regimen during the study and for up to 30 days following discontinuation of treatment.
4. Ability to participate in the study based on overall health of the patient and disease prognosis, as applicable, in the opinion of the Investigator; and able to comply with all requirements of the protocol, including completion of study questionnaires.

Exclusion Criteria:

Individuals who met any of the exclusion criteria in the original protocol or those listed below are not eligible to participate in the study:

1. Epilepsy and currently on medication.
2. Uncontrolled asthma.
3. Concomitant use with sultopride.
4. Concomitant use with medicinal products with a narrow therapeutic window.
5. Concomitant use with medicinal products with a known to cause QTc prolongation.
6. Clinically significant abnormalities in 12 lead ECG, in the opinion of the Investigator.
7. Subjects with congenital QT syndromes.
8. Breastfeeding or pregnant at Screening or planning to become pregnant at any time during the study.
9. Intolerable amifampridine-related side effects
10. Treatment with an investigational drug (other than amifampridine) or device while participating in this study.
11. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confound the assessment of the patient.
12. History of drug allergy to any pyridine-containing substances or any amifampridine excipient(s).

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Maggi, MD, Principal Investigator — Carlo Besta Institute, Milan, Italy
Locations (1):
- Neurological Institute Carlo Besta, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amifampridine Phosphate
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amifampridine Phosphate
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants] — Male or female between the ages of 6 and 50 years and who had completed the SMA-001. This is part of the eligibility criteria.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 13
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 6
  Serbia | 7
Height [Mean (Full Range); unit: CM] | 171.9 [163 to 187]
Weight [Mean (Full Range); unit: Kg] | 67.1 [53 to 86]
BMI [Mean (Full Range); unit: kg/m^2] | 22.7 [16.7 to 28.4]

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety and Tolerability of Amifampridine
Description: Number of subjects with treatment emergent adverse events (TEAE).
Time Frame: 18 months
Population: TEAE = any AE started at or after the first dose of drug for the current Long-Term Study.
Measure: Count of Participants; unit: Participants
Arm/Group | Amifampridine Phosphate
Number analyzed (Participants) | 13
Participants | 5
Statistical Analysis 1: Comparison: Amifampridine Phosphate; Test type: Other; percentage = 38.5

2. Secondary Outcome: To Assess the Clinical Efficacy of Amifampridine Phosphate Over Time in Patients With SMA Type 3 Based on Changes in Quality of Life (QoL).
Description: Quality of life (QoL): the Individualized Quality of Life for neuromuscular disease (INQoL) or the Pediatric Quality of Life (PEDSQLTM) was used for adult or pediatric patients, respectively. Since there were no pediatric patients, none of the patients completed the PEDSQL.
  The INQol evaluated weakness, pain, fatigue, double vision, muscle locking, droopy eyelids, swallowing difficulties, activities, social relationships, emotions and body image. Each of these areas were measured in four categories as follows: 1- Incidence (0= No, 1 =Yes), 2-Severity (0= None to 7 = extreme), 3- Impact - (0= None to 6 = extreme) and 4-Importance (0= None to 6 = extreme). The numbers were summative and are input to the QOL calculation, which is a percentage of severity on a scale of 0-100. The mean value was taken across this population. The higher scores were a worse outcome.
Time Frame: Screening to end of study.
Population: 11 patients completed the screening Quality of Life Score and only 9 patients completed the EOS Quality of Life Score .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amifampridine Phosphate
Number analyzed (Participants) | 11
score on a scale
  screening | 33.737 (17.677)
  End of Study: number analyzed (Participants) | 09
  End of Study | 39.012 (14.337)

ADVERSE EVENTS:
Time Frame: 27 months
Description: The reporting period for SAEs began after obtaining informed consent and continued through 4 weeks after the last visit. A treatment emergent adverse event (TEAE) was defined as any AE that started at or after the first dose of study drug for the long-term study.
Arm/Group | Amifampridine Phosphate
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amifampridine Phosphate (N=13)
Intellectual Disability (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amifampridine Phosphate (N=13)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2)
HYPERPYREXIA (General disorders) | 2 (2)
FEELING HOT (General disorders) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1)
MALAISE (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
POST LUMBAR PUNCTURE SYNDROME (General disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The results of efficacy are limited to the assessment of quality of life using the INQoL. The premature interruption of the study determined that few patients had available data of INQoL from Month 6 onwards.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: original protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03819660/Prot_000.pdf
  • Study Protocol: Amendment 1 (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03819660/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03819660/SAP_002.pdf